CLINICAL TRIAL: NCT03690791
Title: A Randomised, Double-blind, Single-centre Study on the Safety, Tolerability and Efficacy of Cannabis Based Medicine Extract (MediCabilis CBD Oil) in Slowing the Disease Progression in Amyotrophic Lateral Sclerosis or Motor Neurone Disease Patients
Brief Title: Efficacy of Cannabinoids in Amyotrophic Lateral Sclerosis or Motor Neurone Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: Bod Australia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCMR0001
Record Dates: First submitted 2018-09-13; First posted 2018-10-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MediCabilis CBD Oil (Active Comparator)
  Interventions: Drug: MediCabilis CBD Oil
- Placebo Oil (Placebo Comparator)
  Interventions: Drug: Placebo Oil

INTERVENTIONS:
Drug: MediCabilis CBD Oil — 50 mg of CBD: <2mg of THC in one ml. The cannabis oil consists of CBD extract in MCT oil.
  Arms: MediCabilis CBD Oil
Drug: Placebo Oil — Placebo will contain only hemp seed oil.
  Arms: Placebo Oil

SUMMARY:
This is a randomised, double-blind, placebo controlled study on a cannabis-based medicine extract (MediCabilis CBD Oil), in patients with Amyotrophic Lateral Sclerosis or Motor Neurone Disease. Participants will be randomised in a 1:1 ratio to receive MediCabilis CBD Oil or placebo oil. The treatment duration is 6 months with one-month safety follow up. Participants will be checked every month either face to face or via telephone and will be assessed to collect data for study objectives such as ALSFRS-R, Forced Vital Capacity, pain and spasticity score, and quality of life. Thirty (30) participants will be randomised.

ELIGIBILITY:
Inclusion Criteria:

1. Affected by ALS/MND, either of definite or probable according to the El Escorial revised criteria
2. Can provide written informed consent
3. Able and willing to comply with all study requirement
4. Male or female, ages 25-80 years old
5. Onset of first symptom within the last 2 years
6. Forced Vital Capacity (FVC) of at least 60% on baseline

Exclusion Criteria:

1. Participants who are bedridden
2. Have used or taken cannabis or cannabinoid-based medications within 30 days of study entry
3. History of any psychiatric disorder other than depression associated with their underlying condition including immediate family history of schizophrenia
4. Heavy consumption of alcohol or use of illicit drug
5. Hypersensitivity to cannabinoids or any of the excipients
6. Any of the following: eGFR <30 mL/min/1.73m2, ejection fraction <35%, or ASL and ALT >5 X ULN
7. Unwillingness of a female participant of child bearing potential, or their partner, to use effective contraception during the study and 30 days thereafter
8. Pregnant, lactating mother or female participant planning pregnancy during the course of the study and for 30 days thereafter
9. Received any investigational drug or medical device within 30 days prior randomisation
10. Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
11. Inability to cooperate with the study procedures
12. Unwilling to stop driving vehicle or operating dangerous machinery whilst on study drug.
13. Close affiliation with the study team, e.g. close relative of the investigator

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Difference in mean ALS Functional Rating Scale-Revised (ALSFRS-R) total score between groups at end of treatment (Total score: min 0- max 48) [efficacy] | Baseline to Day 180
  Change from baseline in ALS functional rating total scores on the ALSFRS-R at 24 weeks. Total score ranges from 0 to 48. Higher value represents better outcome.
Difference in mean Forced Vital Capacity (FVC) volume between groups at end of treatment [efficacy] | Baseline to Day 180
  Change from baseline in Forced Vital Capacity volume on the Lung Function Test at 24 weeks

SECONDARY OUTCOMES:
Nature and number of adverse events [safety and tolerability] | Baseline to Day 180
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 at 24 weeks
Difference in mean Numeric Rating Scale for spasticity total score between groups at end of treatment (Scores 0-100) | Baseline to Day 180
  Change from baseline in spasticity total score on the Numeric Rating Scale for spasticity at 24 weeks. Total score ranges from 0 to 100. Higher values represent better outcome.
Difference in mean Numeric Rating Scale for pain total score between groups at end of treatment (Total score min:1-max:100) | Baseline to Day 180
  Change from baseline in pain total score on the Numeric Rating Scale for pain at 24 weeks. Total score ranges from 0 to 100. Higher value represents better outcome.
Difference in mean Percentage of Total Weight Loss score between groups at end of treatment (Percentage score min: 0- max: 100) | Baseline to Day 180
  Change from baseline in weight loss on the Percentage of Total Weight Loss at 24 weeks. Percentage ranges from 0 to 100. Higher value represents better outcome.
Difference in mean ALS Specific Quality of Life- Revised (ALSSQOL-R) total score between groups at end of treatment (Total score min:0- max:460) | Baseline to Day 180
  Change from baseline in quality of life total score on the ALS Specific Quality of Life- Revised (ALSSQOL-R) score at 24 weeks. Total score ranges from 0 to 460. Higher score represent better outcome.

OTHER OUTCOMES:
Difference in mean Edinburgh Cognitive and Behavioural ALS Screen (ECAS) total score between groups at end of treatment (Score 0-136) | Baseline to Day 180
  Change from baseline in quality of life total score on the ALS Specific Quality of Life- Revised (ALSSQOL-R) total score at 24 weeks. Total score ranges from 0 to 100. Higher score represent better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Gold Coast Hospital and Health Service, Gold Coast, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the Australian Government Data Sharing Policy, the NHMRC Open Access Policy and the Clinical Trials Registration and Results Information Submission rule.
  Additional data can be requested from the authors. However, the decision to disclose data is solely based from authors' discretion and funding agency.

REFERENCES:
- [Derived] Urbi B, Broadley S, Bedlack R, Russo E, Sabet A. Study protocol for a randomised, double-blind, placebo-controlled study evaluating the Efficacy of cannabis-based Medicine Extract in slowing the disease pRogression of Amyotrophic Lateral sclerosis or motor neurone Disease: the EMERALD trial. BMJ Open. 2019 Nov 11;9(11):e029449. doi: 10.1136/bmjopen-2019-029449. PMID 31719072